CLINICAL TRIAL: NCT05484635
Title: Mesh Removal Versus No Mesh Removal for Chronic Groin Pain After Minimally Invasive Inguinal Hernia Repair: A Randomized Controlled Trial
Brief Title: Mesh Removal Versus No Mesh Removal for Chronic Groin Pain After Inguinal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Krpata (Other)
Responsible Party: Sponsor-Investigator, David Krpata, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-411
Record Dates: First submitted 2022-07-26; First posted 2022-08-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Chronic Groin Pain; Hernia, Inguinal
Keywords: Chronic groin pain; Hernia, Inguinal; Chronic pain groin
MeSH Terms: conditions — Hernia, Inguinal | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diagnostic laparoscopy (Active Comparator): Minimally invasive incisions will be made, and a diagnostic laparoscopy will be performed. The surgeon will evaluate the mesh configuration, ensuring proper positioning, perform adhesiolysis if indicated for bowel involvement with the mesh and assess the abdomen for alternative sources of chronic pain.
  Interventions: Procedure: Diagnostic laparoscopy
- Laparoscopic mesh removal (Experimental): Minimally invasive incisions will be made, and a diagnostic laparoscopy will be performed. The surgeon will evaluate the mesh configuration, ensuring proper positioning, perform adhesiolysis if indicated for bowel involvement with the mesh and assess the abdomen for alternative sources of chronic pain. If randomized to mesh removal, laparoscopic or robotic preperitoneal mesh removal.
  Interventions: Procedure: Diagnostic laparoscopy and inguinal mesh removal

INTERVENTIONS:
Procedure: Diagnostic laparoscopy and inguinal mesh removal — Surgical examination and treatment of groin pain following inguinal hernia surgery by surgical exploration with a laparoscope or removal of mesh laparoscopically
  Arms: Laparoscopic mesh removal
Procedure: Diagnostic laparoscopy — Surgical examination through laparoscopy without removal of mesh
  Arms: Diagnostic laparoscopy

SUMMARY:
This study is evaluating the management of chronic post-operative inguinal hernia pain and the impact of hernia mesh removal after previous minimally invasive inguinal hernia repairs.

The study aims are to evaluate the change in chronic (>6 months), nociceptive, postoperative inguinal pain after mesh removal compared to no mesh removal in patients who have previously undergone minimally invasive inguinal hernia repair with pre-peritoneal mesh.

DETAILED DESCRIPTION:
This is a double-blinded, parallel (1:1) group, randomized-controlled, superiority trial. Patients will be blinded to their treatment allocation and will understand that by entering the study, they may receive diagnostic laparoscopy only in which case their mesh will not be removed. However, they will be allowed to consider crossing over to the mesh removal group 6 months or later after surgery if they do not have adequate pain relief. Patients will receive written and oral descriptions of the trial and will be provided time to review written documentation in private. Written and oral consent will be obtained, and patients will understand that their participation is voluntary and refusal to participate will not affect future medical care. Patients may also withdraw from the trial at any point throughout the study period.

The Cleveland Clinic Center for Abdominal Core Health, a center within the Digestive Disease and Surgery Institute (DDSI), at Cleveland Clinic Foundation Main Campus in Cleveland, Ohio is the hosting department for this study. Cleveland Clinic - Hillcrest Hospital in Mayfield Heights, Ohio will also be a participating center in this study. Fellowship-trained surgeons with expertise in complex abdominal wall reconstruction and mesh removal will perform the operations. If enrollment fails to meet necessary accrual size within the study timeframe, additional centers may be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* CPIP lasting > 6 months after laparoscopic or robotic inguinal hernia repair with pre-peritoneal mesh
* Must exhibit 1 or more of the following characteristics of nociceptive pain:

History:

* Pain while sitting in a chair for prolonged periods of time with relief when extending the hip or lying supine to straighten the leg
* Severe pain when crossing the affected leg over the contralateral leg
* "Foreign body sensation" or "tightness" in the groin

Exam:

-Diffuse tenderness with deep palpation along the inguinal ligament (over the mesh)

Somatosensory mapping:

* Does not have a maximum trigger point for pain
* Lacks characteristics of neuropathic pain (sharp, burning, shooting, paresthesias, allodynia, hyperalgesia, etc.)

  * Moderate to severe pain [4-10] when moving from supine to standing on NRS

Exclusion Criteria:

* No characteristics of nociceptive groin pain
* Zero or mild pain [0-3] when moving from supine to standing on NRS
* Recurrent inguinal hernia detected on clinical exam
* Large, femoral, direct or indirect inguinal hernia (F2-3, M2-3, L2-3) on diagnostic laparoscopy as defined by European Hernia Society (EHS) classification
* Prior open (anterior) approach to inguinal hernia repair (i.e. Lichtenstein)
* Prior mesh plugs or Prolene Hernia Systems
* History of prostatectomy or vascular procedures in the pelvis or groin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS-11) | Change in NRS-11 scores will be measured from baseline to 6 months after surgery for both groups.
  NRS-11 is a validated, 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) and is commonly used to measure Chronic Post-operative Inguinal Pain (CPIP). NRS-11 categorizes pain as none [0], mild [1-3], moderate [4-6], and severe [7-10]. Patients will be asked to select the single number that best represents their groin pain intensity when moving from a supine to standing position.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 3-months and 6-months
  VAS is validated and consists of a 100 mm horizontal line anchored by two descriptors indicating the extremes: 0 (no pain) and 100 (worst pain imaginable).
Activities Assessment Scale (AAS) | Baseline, 3-months and 6-months
  AAS is a 13-item, validated tool measuring physical impairment due to chronic groin pain. AAS scores are converted to a range of 0-100, with higher values indicating better functional ability.
EuroQOL (EQ-5D-5L) questionnaire | Baseline, 3-months and 6-months
  EQ-5D-5L is a validated tool evaluating 5 dimensions of health using 5 severity descriptors and includes a visual analog scale labeled from 0 to 100 to quantitatively measure overall health status. The larger the number the better the outcome.
Numerical Rating Scale (NRS-11) | Baseline NRS-11 scores will be measured and compared to scores at 3 months after surgery for both groups.
  NRS-11 is a validated, 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) and is commonly used to measure Chronic Post-operative Inguinal Pain (CPIP). NRS-11 categorizes pain as none [0], mild [1-3], moderate [4-6], and severe [7-10]. Patients will be asked to select the single number that best represents their groin pain intensity when moving from a supine to standing position.

CONTACTS AND LOCATIONS:
Overall Officials: David Krpata, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided